CLINICAL TRIAL: NCT01847144
Title: MASTERMIND - Understanding Individual Variation in Treatment Response in Type 2
Brief Title: MASTERMIND - Understanding Individual Variation in Treatment Response in Type 2 Diabetes
Acronym: Mastermind
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CRF111; MR/K005707/1 (Other Grant/Funding Number: MRC grant reference)
Record Dates: First submitted 2013-03-13; First posted 2013-05-06 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gliclazide; Dipeptidyl-Peptidase IV Inhibitors; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gliclazide - Sitagliptin (Active Comparator): Gliclazide 80mg OD and Sitagliptin 100mg OD
  Interventions: Drug: Gliclazide 80mg OD
- Sitagliptin - Gliclazide (Active Comparator): Gliclazide 80mg OD and Sitagliptin 100mg OD
  Interventions: Drug: Sitagliptin 100mg OD

INTERVENTIONS:
Drug: Gliclazide 80mg OD — Gliclazide 80mg OD (DPP-IV inhibitor) - for 4 weeks duration followed by a 2 week wash-out period.
  Other Names: DPP-IV inhibitor
  Arms: Gliclazide - Sitagliptin
Drug: Sitagliptin 100mg OD — Sitagliptin 100mg OD (sulphonylurea)- for 4 weeks duration followed by a 2 week wash-out period.
  Other Names: sulphonylurea OD
  Arms: Sitagliptin - Gliclazide

SUMMARY:
Response to treatment in Type 2 Diabetes is highly variable; the same medicine may have little effect in one person but a large effect in another. Understanding mechanisms of altered response to treatment could aid treatment selection and assist the design of new medications with lower nonresponse rates.

This study will examine the physiological mechanisms and potential clinical/biomarker predictors of altered response to sulphonylurea and DPPIV inhibitor glucose lowering medication and answer fundamental methodological questions for the future study of variation in treatment response in Type 2 Diabetes. Participants will withdraw sulphonylurea therapy for up to 2 weeks with assessment of baseline characteristics and glycaemic response. Participants will then enter an optional extension where they receive sulphonylurea or DPPIV inhibitor therapy in crossover fashion.

DETAILED DESCRIPTION:
Participants will withdraw sulphonylurea therapy for up to 2 weeks (part 1) followed by an optional cross-over extension (part 2)where they are randomized to 4 weeks of treatment with Gliclazide (DPP-IV thera) or Sitagliptin (sulphonylurea), followed by 4 weeks of the second treatment with a 2 week wash-out period in between.

Part 1 will allow assessment of response rates to long standing sulphonylurea treatment in clinical practice and potential predictors of this, as well as whether a very brief period (1 week) of treatment withdrawal is a valid assessment of an individual's response to therapy. Part 2 will allow comparison of the approach in part one with response to the same treatment in a trial setting and will allow assessment on whether response is consistent across therapies with different mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <80
* Clinical diagnosis of Type 2 Diabetes
* Currently treated with sulphonylurea tablets
* No change in diabetes treatment (new treatments or dose change) within last 3 months
* Last HbA1c (taken within last 12 months) of ≥42 mmol/mol and ≤75 mmol/mol (6-9%)
* Able and willing to monitor home blood glucose
* Able and willing to give informed consent

Exclusion Criteria:

* Current treatment includes: insulin, GLP-1 agonists, DPP-IV inhibitors, glinides
* Renal impairment (eGFR <30 ml/min/1.73m2)
* Active infection (any infection requiring antibiotics at present)
* Recent (within 3 months) surgery or planned surgery
* Cardiovascular disease (angina, myocardial infarction, stroke, transient ischemic episode) occurring within the previous 3 months
* Previous history of pancreatitis
* Pregnant, breastfeeding or planning a pregnancy over the study period
* Unable/unwilling to monitor home blood glucose

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in fasting glucose | 4 weeks post treatment change
  Change in fasting glucose from 0 to 4 weeks post treatment change.

SECONDARY OUTCOMES:
Additional changes in biochemical results | 4 weeks
  Secondary outcome measures will include change in glycosylated albumin, HbA1c, home glucose day profile and mixed meal area under the curve glucose

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, FRCP, DM, BM, Principal Investigator — University of Exeter
Locations (1):
- NIHR Exeter Clinical Research Facility, Royal Devon & Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom